CLINICAL TRIAL: NCT06657820
Title: Optical Brain Pulse Monitor: Validation Of Cerebral Oximetry Monitoring (OBPM: VOCOM) Study.
Brief Title: Optical Brain Pulse Monitor: Validation Of Cerebral Oximetry Monitoring (OBPM:VOCOM) Study.
Acronym: OBPM:VOCOM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The decision was made to withdraw this study prior to recruitment to make further changes to the investigational device.
Sponsor: Elliot Teo (Industry)
Collaborators: Duke University Hospital, USA (Unknown)
Responsible Party: Sponsor-Investigator, Elliot Teo, Clinical Research Manager, Cyban Pty Ltd
Organization: Cyban Pty Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00116391
Record Dates: First submitted 2024-10-15; First posted 2024-10-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-09

CONDITIONS: Hypoxia
Keywords: Cerebral Oximetry; Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Subject will undergo a graduated desaturation protocol beginning at 100%, then 99%, then descending in 3% increments to a final target of 66%. Arterial and venous jugular bulb co-oximetry measurements will be taken at each saturation plateau yielding a total of 13 paired samples per subject. The weighted average of the SaO2 and the SvO2 will be compared against the Cyban Cerebral Oximeter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Desaturation (Experimental): A central venous catheter will be placed in the right internal jugular vein and the catheter tip advanced retrograde to lie at the level of the jugular bulb. An arterial catheter will be placed in the forearm. A dedicated breathing circuit will be used to reduce the alveolar oxygen tension (PAO2) in stepwise fashion to produce a controlled oxygen desaturation sequence. The dedicated breathing circuit will be used to maintain the alveolar carbon dioxide tension (PACO2) at normocapnic value of 40 mmHg. At each step once steady state conditions are achieved, serial paired arterial and jugular bulb venous samples will be drawn. The blood gas samples will be analyzed by Radiometer ABL90 Flex CO-oximeter.
  Interventions: Procedure: Hypoxia in healthy individuals; Device: Cerebral Oximetry; Diagnostic Test: Blood Gas Sampling

INTERVENTIONS:
Procedure: Hypoxia in healthy individuals — The subject will undergo a graduated desaturation procedure. Arterial saturation targets are as follows:
  1. 100%
  2. 99%
  3. 96%
  4. 93%
  5. 90%
  6. 87%
  7. 84%
  8. 81%
  9. 78%
  10. 75%
  11. 72%
  12. 69%
  13. 99%
Device: Cerebral Oximetry — Each subject will be continuously monitored with the cerebral oximetry device throughout the desaturation procedure.
Diagnostic Test: Blood Gas Sampling — At each arterial saturation plateau venous and arterial blood gas measurements will be taken from the jugular bulb, and the radial artery respectively.

SUMMARY:
The purpose of this study is to calibrate and validate a cerebral oximeter product from Cyban Pty. Ltd. The study will involve comparing cerebral oximeter signals against reference arterial and jugular bulb blood gas measures.

DETAILED DESCRIPTION:
The primary objective of the study is to measure the absolute and relative accuracy of the StO2 device by comparing the NIRS-derived brain tissue oxygen saturation with blood-referenced CO-oximeter oxygen saturation values. The CO-oximeter oxygen saturation values from paired arterial and jugular bulb blood samples are combined into a weighted-equation to derive the reference SavO2. Accuracy is reported over a range of oxygen saturations with study subjects exposed to a controlled oxygen desaturation with serial sampling of paired arterial and internal jugular venous blood gas samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female subjects between the ages of 18 to 45 years;
* Completion of a health screening for a medical history by a licensed physician, nurse practitioner, or physician assistant;
* Minimum weight 40kg;
* BMI within range 18.0 - 35.0;
* Assigned American Society of Anesthesiologists (ASA) Physical Status 1 by Principal Investigator or delegate

Exclusion Criteria:

* Prior or known allergies to lidocaine (or similar pharmacologic agents, e.g., Novocain) [self- reported];
* Prior known severe allergies to medical grade adhesive/tape (Band-Aid) [self-reported];
* Taking any medication other than birth control[self-reported];
* Is currently participating in, or has recently participated in (discontinued within 30 days prior to the hypoxia procedure for this study) in an investigational drug, device, or biologic study [self- reported];
* Has a negative Allen's Test to confirm non-patency of the collateral artery [clinical assessment by PI or delegate];
* Has made a whole blood donation or has had at least 450 ml of blood drawn within 8 weeks prior to the study procedure [self-reported];
* Is female with a positive pregnancy test [serum or urine], or is female and is unwilling to use effective birth control between the time of screening and study procedure or is breast feeding;
* Has anemia [lab values specific for gender];
* Has heparin allergy
* Has a history of sickle cell trait or thalassemia [self-reported];
* Has an abnormal hemoglobin electrophoresis result [lab measurement];
* Has a positive urine cotinine test or urine drug screen or oral ethanol test;
* Has a room air saturation less than 95% by pulse oximetry [measurement by PI or delegate]
* Has a clinically significant abnormal EKG [assessment by PI or delegate];
* Has a clinically significant abnormal pulmonary function test via spirometry [assessment by PI or delegate];
* Has a COHb greater than 3%, or MetHb greater than 2% [measured by venous blood sample co- oximetry].
* Students and Employees under the direct supervision of PI or Sub-I.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-06 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy by Average Root Mean Squared Error | 6 months
  The Accuracy by Root Mean Square Difference (ARMS) will be used to evaluate accuracy of the investigational device StO2 compared with the blood-referenced SavO2
Bland-Altman Agreement Analysis | 6 months
  A Bland-Altman (BA) analysis will be conducted on the difference (D) and mean (A) of StO2, SavO2, where
  * D = StO2 - SavO2
  * A = (StO2 + SavO2) / 2
  The following statistics will be presented:
  * Bias and its 95% confidence interval (CI)
  * Standard deviation of bias (sum of between and within subject variance components)
  * Lower and upper 95% limit of agreement (LoA) and their 95% CI

SECONDARY OUTCOMES:
Concordance Correlation Coefficient | 6 months
  The concordance correlation coefficient (CCC) method is used to measure the agreement between of two devices. CCC could have values from -1 to 1, with values near 1 indicating strong concordance between the two devices, values near -1 indicating strong discordance, and values near zero indicating no concordance.
Passing-Bablok Regression Analysis | 6 months
  Passing-Bablok regression is used to compare measurements from different devices, and is a robust nonparametric regression method that does not make assumptions about the distribution of the expected values or the error terms in the model. The 95% CI for the intercept and slope will be estimated from the regression.
Linear Mixed Model Regression Analysis | 6 months
  A random effects linear mixed model will be used to regress StO2 on SavO2. Subject will be included as a random effect in the model to account for the correlation of repeated measures within the same subject.
Subgroup Analysis of Agreement | 6 months
  Bland-Altman analyses will be generated for subgroups to assess the two device agreement among different subgroups. A forest plot will used to present the results. The following subgroups will be considered.
  * Restricted oxygen desaturation range: 50% ≤ reference SavO2 ≤ 75%
  * Oxygen desaturation steps as measured by SpO2 (13 steps)
  * Fitzpatrick score group
  * Sex
  * Race

OTHER OUTCOMES:
Safety Analyses | 6 months
  All safety analyses will be conducted on the Safety Population. No inferential statistical testing will be performed for safety variables.
  Any reported adverse events, safety observations, and adverse device deficiencies will be listed in a separate by participant data listing.

CONTACTS AND LOCATIONS:
Overall Officials: David B Macleod, M.B.B.S, Principal Investigator — Human Pharmacology and Physiology Lab, Department of Anesthesiology, Duke University Medical Center, Durham, North Carolina, USA

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.